CLINICAL TRIAL: NCT00780741
Title: A Randomized Trial Comparing Immediate Probing in an Office Setting With Deferred Probing in a Facility Setting for Treatment of Nasolacrimal Duct Obstruction in Children 6 to <10 Months Old
Brief Title: Immediate Office Probing vs Deferred Facility Probing for Nasolacrimal Duct Obstruction in Children 6 to <10 Months Old
Acronym: NLD3
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Jaeb Center for Health Research (Other)
Collaborators: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NEI-142; 2U10EY011751 (NIH)
Record Dates: First submitted 2008-10-27; First posted 2008-10-28 (Estimated); Results first posted 2012-11-12 (Estimated); Last update posted 2016-06-24 (Estimated); Status verified 2016-05

CONDITIONS: Nasolacrimal Duct Obstruction
Keywords: Nasolacrimal duct obstruction; Simple probing
MeSH Terms: conditions — Lacrimal Duct Obstruction

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Immediate Office Probing (Active Comparator): Probing to be performed in the office setting using topical anesthesia and infant restraint. Probing to be performed either the same day as randomization or within two weeks.
  Interventions: Procedure: Immediate Office Probing
- Deferred Facility Probing (Active Comparator): Probing to be performed in a surgical facility under general anesthesia within four weeks after completion of the 26-week visit if any of the clinical signs persist.
  Interventions: Procedure: Deferred Facility Probing

INTERVENTIONS:
Procedure: Immediate Office Probing — Nasolacrimal duct probing in an office setting with topical anesthesia and restraint of the infant.
  Arms: Immediate Office Probing
Procedure: Deferred Facility Probing — Nasolacrimal duct probing performed under general anesthesia in a hospital outpatient surgery center or an ambulatory surgery center.
  Arms: Deferred Facility Probing

SUMMARY:
The purpose of this study is:

To determine the cost-effectiveness of treating NLDO using immediate office probing compared with deferred probing in a facility setting. As part of the primary objective, the study will determine the proportion of eyes experiencing spontaneous resolution among subjects randomized to the deferred probing group.

The secondary objectives are:

1. To determine the success proportion for eyes undergoing immediate office probing as an initial procedure.
2. To determine the success proportion for eyes undergoing deferred facility probing as an initial procedure.

DETAILED DESCRIPTION:
Nasolacrimal duct obstruction (NLDO) is a common ocular condition in the first year of life. Many cases will resolve spontaneously or with massage. Many studies of primary treatment of NLDO have been reported, however these case series have largely been retrospective, uncontrolled, and conducted in single centers. The substantial uncertainty regarding an estimate of spontaneous resolution is a primary reason for conducting the current study.

Probing is the most widely-used initial treatment for NLDO in infancy. Our group recently completed a prospective observational study which found a 78% success proportion of probing among children aged 6 to <12 months. Other estimates of the success rate for probing vary between 69% and 92%.

Two differing approaches to nasolacrimal probing have been most often been used: (1) immediate office probing (early probing - generally soon after 6 months of age) and (2) medical management (episodic antibiotic eye drops with massage of the lacrimal sac) until 9-13 months of age followed by probing under general anesthesia or conscious sedation (deferred probing). The advantages of early probing are the avoidance of general anesthesia or conscious sedation, immediate resolution of symptoms, fewer physician visits, fewer antibiotic prescriptions, lesser cost per procedure, and possible prevention of fibrosis from inflammation in the nasolacrimal duct. The advantages of deferred probing include more subject comfort with the procedure and possible avoidance of a surgical procedure completely.

The optimal approach to the management of NLDO in the first year of life remains uncertain. Our prospective observational data suggest a slightly reduced chance of success with immediate office probing (75% for office probing, 80% for facility probing), however, immediate office probing may be more cost-effective even if the proportion with success is lower. For a subject undergoing a single operation, immediate office probing is less expensive than deferred probing in a facility because there is no fee for anesthesia, the facility, or for medications prescribed during the pre-operative observation period. Some portion of this lower cost would be offset however by the additional cost of a second procedure if the initial office probing is not successful. Deferred facility probing is more expensive per procedure; however, the overall costs are reduced by the number of children whose NLDO spontaneously resolves while waiting to perform the procedure in a facility.

The study is a randomized clinical trial which aims to determine the cost-effectiveness of treating NLDO using immediate office probing compared with deferred probing in a facility setting. As part of the primary objective, the study will determine the proportion of eyes experiencing spontaneous resolution among subjects randomized to the deferred probing group.

ELIGIBILITY:
Inclusion Criteria:

* Age 6 to <10 months
* Onset of NLDO symptoms and/or signs prior to 6 months chronological age in study eye(s)
* Presence in study eye(s) of epiphora, increased tear film, and/or mucous discharge in the absence of an upper respiratory infection or an ocular surface irritation that investigator believes is due to NLDO
* At least one open punctum present in study eye(s)

A history of NLDO treatment with lacrimal massage, topical antibiotics or steroids, or systemic antibiotics is permitted.

Exclusion Criteria:

* History of nasolacrimal duct surgery including probing, nasolacrimal intubation, balloon catheter dilation, or dacryocystorhinostomy in study eye(s) History of trauma to the lacrimal drainage system of the study eye(s)
* Glaucoma in study eye(s)
* Corneal surface disease in study eye(s)
* Microphthalmia in study eye(s)
* Down Syndrome
* Craniosynostosis
* Goldenhar sequence
* Clefting syndromes
* Hemifacial microsomia
* Midline facial anomalies

Ages: 6 Months to 10 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 220 (Actual)
Dates: Start 2008-10; Primary Completion 2011-11 (Actual); Study Completion 2012-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Katherine A. Lee, M.D., Ph.D., Study Chair — Intermountain Eye Centers
Locations (1):
- Intermountain Eye Centers, Boise, Idaho, United States

REFERENCES:
- [Background] Pediatric Eye Disease Investigator Group. Resolution of congenital nasolacrimal duct obstruction with nonsurgical management. Arch Ophthalmol. 2012 Jun;130(6):730-4. doi: 10.1001/archophthalmol.2012.454. PMID 22801833
- [Background] Lee KA, Chandler DL, Repka MX, Melia M, Beck RW, Summers CG, Frick KD, Foster NC, Kraker RT, Atkinson S; PEDIG. A comparison of treatment approaches for bilateral congenital nasolacrimal duct obstruction. Am J Ophthalmol. 2013 Nov;156(5):1045-50. doi: 10.1016/j.ajo.2013.06.014. Epub 2013 Aug 15. PMID 23954210
- [Background] Miller AM, Chandler DL, Repka MX, Hoover DL, Lee KA, Melia M, Rychwalski PJ, Silbert DI; Pediatric Eye Disease Investigator Group; Beck RW, Crouch ER 3rd, Donahue S, Holmes JM, Quinn GE, Sala NA, Schloff S, Wallace DK, Foster NC, Frick KD, Golden RP, Lambert SR, Tien DR, Weakley DR Jr. Office probing for treatment of nasolacrimal duct obstruction in infants. J AAPOS. 2014 Feb;18(1):26-30. doi: 10.1016/j.jaapos.2013.10.016. PMID 24568978
- [Result] Pediatric Eye Disease Investigator Group. A randomized trial comparing the cost-effectiveness of 2 approaches for treating unilateral nasolacrimal duct obstruction. Arch Ophthalmol. 2012 Dec;130(12):1525-33. doi: 10.1001/archophthalmol.2012.2853. PMID 23229693
- See also: PubMed Abstract — https://www.ncbi.nlm.nih.gov/pubmed/23229693
- See also: PubMed Central HHS Public Access - Full Text — http://www.ncbi.nlm.nih.gov/pmc/articles/PMC3537230/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Between November 2008 and September 2010, 163 participants with unilateral nasolacrimal duct obstruction (NLDO) were enrolled at 22 clinical centers.
  During the same period, 57 participants were recruited with bilateral nasolacrimal duct obstruction (NLDO), however, these participants are not included in the analyses reported herein.
Groups:
- Immediate Office Probing - Participants With Unilateral NLDO: Probing to be performed in the office setting using topical anesthesia and infant restraint. Probing to be performed either the same day as randomization or within two weeks. Limited to participants with unilateral nasolacrimal duct obstruction (NLDO).
- Deferred Facility Probing - Participants With Unilateral NLDO: Probing to be performed in a surgical facility under general anesthesia within four weeks after completion of the 26-week visit if any of the clinical signs persist. Limited to participants with unilateral nasolacrimal duct obstruction (NLDO).
Period: Overall Study
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO | Deferred Facility Probing - Participants With Unilateral NLDO
Started | 82 (randomized) | 81 (randomized)
6-Month Visit | 73 (6 months (±2 weeks) timed from randomization) | 67 (6 months (±2 weeks) timed from randomization)
Completed | 75 (18 months of age (±4 weeks)) | 71 (18 months of age (±4 weeks))
Not Completed | 7 | 10

BASELINE CHARACTERISTICS:
Groups:
- Immediate Office Probing - Participants With Unilateral NLDO: Probing to be performed in the office either the same day as randomization or within two weeks. Limited to participants with unilateral nasolacrimal duct obstruction (NLDO).
- Deferred Facility Probing - Participants With Unilateral NLDO: Probing to be performed in a facility within four weeks after completion of the 26-week visit if any of the clinical signs persist. Limited to participants with unilateral nasolacrimal duct obstruction (NLDO).
- Total: Total of all reporting groups
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO | Deferred Facility Probing - Participants With Unilateral NLDO | Total
Number analyzed (Participants) | 82 | 81 | 163
Age, Continuous [Mean (Standard Deviation); unit: months] | 7.6 (1.2) | 7.8 (1.3) | 7.7 (1.2)
Age, Customized [Number; unit: participants]
  6 to <7 months | 25 | 27 | 52
  7 to <8 months | 28 | 20 | 48
  8 to <9 months | 15 | 13 | 28
  9 to <10 months | 14 | 21 | 35
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 32 | 42 | 74
  Male | 50 | 39 | 89
Race/Ethnicity, Customized [Number; unit: participants]
  White | 68 | 66 | 134
  African American | 3 | 6 | 9
  Hispanic or Latino | 10 | 7 | 17
  Asian | 1 | 1 | 2
  More than one race | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  United States | 82 | 81 | 163
Previous treatment for NLDO [Number; unit: participants]
  Lacrimal massage and topical antibiotics | 39 | 36 | 75
  Lacrimal massage only | 18 | 15 | 33
  Topical antibiotics only | 10 | 14 | 24
  None | 15 | 15 | 30
  Unknown | 0 | 1 | 1
Epiphora [Number; unit: participants]
  Present | 63 | 70 | 133
  Absent | 19 | 11 | 30
Increased tear film [Number; unit: participants]
  Present | 79 | 81 | 160
  Absent | 3 | 0 | 3
Mucous discharge [Number; unit: participants]
  Present | 60 | 63 | 123
  Absent | 22 | 18 | 40

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Treatment Success
Description: Absence of three clinical signs of NLDO (epiphora, increased tear lake, and mucous discharge) upon masked examination at 18 months of age.
Time Frame: 18 months of age
Population: All participants who had unilateral nasolacrimal duct obstruction at baseline and who completed the primary outcome visit at 18 months of age were analyzed. The analysis followed the intent-to-treat principle.
Measure: Number; unit: proportion of participants
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO | Deferred Facility Probing - Participants With Unilateral NLDO
Number analyzed (Participants) | 75 | 71
proportion of participants | 0.92 | 0.82
Statistical Analysis 1: Comparison: Immediate Office Probing - Participants With Unilateral NLDO vs Deferred Facility Probing - Participants With Unilateral NLDO; Test type: Superiority or Other; p = 0.09, Point estimate on mean difference; Bootstrap sampling with replacement (N=10,000) was used to calculate the 95% confidence interval; Mean Difference (Final Values) = 0.10, 95% CI 2-sided [-0.01 to 0.21] — Mean difference calculated as the proportion with success in immediate group minus proportion with success in deferred group. 95% confidence interval obtained using bootstrap sampling with replacement

2. Primary Outcome: Cost of Treatment
Description: Total cost of treatment including the cost of an initial office consultation and all surgeries received (i.e. initial surgeries and reoperations) and medications prescribed for NLDO between randomization and the 18 months of age visit. Estimates of treatment costs were obtained primarily from the 2011 Medicare Fee Schedules.
Time Frame: Randomization to 18 months of age
Population: All participants who had unilateral nasolacrimal duct obstruction at baseline and who completed the visit at 18 months of age were analyzed. The analysis followed the intent to treat principle.
Measure: Mean (Full Range); unit: US dollars
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO | Deferred Facility Probing - Participants With Unilateral NLDO
Number analyzed (Participants) | 75 | 71
US dollars | 562 [141 to 2597] | 701 [141 to 2794]
Statistical Analysis 1: Comparison: Immediate Office Probing - Participants With Unilateral NLDO vs Deferred Facility Probing - Participants With Unilateral NLDO; Test type: Superiority or Other; p = 0.24, Point estimate on mean difference; Bootstrap sampling with replacement (N=10,000) was used to calculate the 95% confidence interval; Mean Difference (Net) = -139, 95% CI 2-sided [-377 to 94] — Mean difference calculated as the average cost in immediate group minus average cost in deferred group. 95% confidence interval obtained using bootstrap sampling with replacement

3. Secondary Outcome: Months of Symptoms of Nasolacrimal Duct Obstruction (NLDO) Between Randomization and 18 Months of Age
Description: Months of NLDO symptoms between randomization and 18 months of age. When resolution of NLDO occurred without surgery, the time of resolution was estimated as the midpoint between randomization and the first time point at which symptoms/signs were reported as absent (i.e. 3-month phone call, 6-month visit, or 18 months of age visit) without a subsequent report of symptoms/signs. For patients who underwent successful surgery, months of symptoms was estimated as months between randomization and the surgery. Patients who had clinical signs present at the 18 month of age visit were considered to have had symptoms present since randomization.
Time Frame: Randomization to 18 months of age.
Population: as for outcome 2
Measure: Mean (Full Range); unit: months of symptoms
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO | Deferred Facility Probing - Participants With Unilateral NLDO
Number analyzed (Participants) | 75 | 71
months of symptoms | 1.8 [0.0 to 12.0] | 4.8 [1.5 to 12.0]
Statistical Analysis 1: Comparison: Immediate Office Probing - Participants With Unilateral NLDO vs Deferred Facility Probing - Participants With Unilateral NLDO; Test type: Superiority or Other; p < 0.0001, Point estimate on mean difference; Bootstrap sampling with replacement (N=10,000) was used to calculate the 95% confidence interval; Mean Difference (Final Values) = -3.0, 95% CI 2-sided [-4.0 to -1.8] — Mean difference calculated as the average months of symptoms in immediate group minus average months of symptoms in deferred group. 95% confidence interval obtained using bootstrap sampling with replacement

4. Secondary Outcome: Proportion of Deferred Facility Probing Group Participants With 6-Month Resolution of NLDO Without Surgery
Description: Absence of three clinical signs of NLDO (epiphora, increased tear lake, and mucous discharge) upon unmasked examination 6 months after randomization. Participants who were operated before the 6-month visit were considered treatment failures.
Time Frame: Randomization to 6 months
Population: All participants who had unilateral nasolacrimal duct obstruction at baseline, who were randomized to the deferred facility probing group, and who completed the 6-month visit (timed from randomization). The analysis followed the intent to treat principle.
Measure: Number (95% Confidence Interval); unit: proportion of participants
Groups:
- Deferred Facility Probing - Participants With Unilateral NLDO: Probing to be performed in a facility within four weeks after completion of the 26-week visit if any of the clinical signs persist.
Arm/Group | Deferred Facility Probing - Participants With Unilateral NLDO
Number analyzed (Participants) | 67
proportion of participants | 0.66 [0.54 to 0.76]

5. Secondary Outcome: Proportion of Participants With Office Probing Success 6 Months After Randomization
Description: The proportion of immediate office group participants whose office probing was successful when assessed 6 months after randomization. Office probing success was defined as absence of three clinical signs of NLDO (epiphora, increased tear lake, and mucous discharge) 6 months after randomization and no reoperation.
Time Frame: Randomization to 6 months
Population: Participants randomized to immediate office probing who underwent office probing.
Measure: Number (95% Confidence Interval); unit: proportion with treatment success
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO
Number analyzed (Participants) | 72
proportion with treatment success | 0.83 [0.73 to 0.90]

ADVERSE EVENTS:
Arm/Group | Immediate Office Probing - Participants With Unilateral NLDO | Deferred Facility Probing - Participants With Unilateral NLDO
Serious Adverse Events (participants affected / at risk) | 0/82 | 0/81
Other Adverse Events (participants affected / at risk) | 0/82 | 0/81

LIMITATIONS AND CAVEATS:
Conclusions not definitive--would need larger sample size.

Participants with bilateral NLDO excluded, so results not generalizable to bilateral cases.

Actual costs may vary by region and payer.

Did not include costs of follow up visits.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No